CLINICAL TRIAL: NCT04701606
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase 2/3 Clinical Trial to Evaluate the Safety and Efficacy of Pyronaridine-artesunate (Artecom®) in COVID-19 Patients
Brief Title: The Safety and Efficacy of Pyronaridine-artesunate (Pyramax® or Artecom®)in COVID-19 Patients
Acronym: PROVIDENCE
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP-PA-COV-203
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Covid19
Keywords: Pyramax; COVID-19; pyronaridine-artesunate; SARS-CoV-2; Artecom
MeSH Terms: conditions — COVID-19 | interventions — pyronaridine tetraphosphate, artesunate drug combination

STUDY DESIGN:
Intervention Model Description: * Stage 1: Single Group (Experimental drug only)
  * Stage 2: Parallel (Placebo control and Experimental drug)
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artecom® (pyronaridine-artesunate) (Experimental): Artecom® is treated orally once a day for 3 consecutive days.
  Interventions: Drug: Artecom® (pyronaridine-artesunate)
- Placebo (Placebo Comparator): Placebo is treated orally once a day for 3 consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Artecom® (pyronaridine-artesunate) — * Participant body weight (Artecom® dose)
  * ≥ 65kg (Artecom® 4 tablets: Pyronaridine 720mg/ Artesunate 240mg)
  * ≥ 45kg and < 65kg (Artecom® 3 tablets: Pyronaridine 540mg/ Artesunate 180mg)
  Other Names: Pyramax® (pyronaridine-artesunate)
  Arms: Artecom® (pyronaridine-artesunate)
Drug: Placebo — * Participant body weight (Placebo dose)
  * ≥ 65kg (Placebo 4 tablets)
  * ≥ 45kg and < 65kg (Placebo 3 tablets)
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, Phase 2/3 study to evaluate the safety and efficacy of pyronaridine-artesunate in participants with corona virus disease 2019 (COVID-19). Pyronaridine-artesunate has been approved in Europe, Asia and Africa under brand name of Pyramax® or Artecom® as a treatment for malaria. The study will be conducted in two stages: open-label (Stage 1) and double-blind (Stage 2).

Up to approximately 402 participants (20 participants in Stage 1 and 382 participants in Stage 2) are planned to be enrolled in the study and will be randomized to receive either Artecom® or matching placebo at a ratio of 1:1 in Stage 2. The dose of Artecom® will be determined by the participant's body weight, according to previously established guidelines.

An independent Drug Safety Monitoring Board (DSMB) will be established to review the safety at regular intervals during the conduct of the trial. The DSMB will be subject to a Charter and will review after 20 participants have been recruited, and thereafter when 191 participants have been recruited.

Ad-hoc DSMB meetings may be held at any time during the study if there are any major safety concerns. A final DSMB will be conducted when all participants have been recruited in the trial.

DETAILED DESCRIPTION:
<Stage 1> In Stage 1, the trial will be conducted in 20 participants for 28 days in a single arm, open-label design. Artecom® will be administered orally once a day for 3 consecutive days. All subjects will be evaluated for efficacy and safety for 28 days.

After the completion of the final participant in Stage 1, the DSMB will review the safety data from Stage 1 and determine whether to proceed to Stage 2.

<Stage 2> In Stage 2, a total of 382 participants will be enrolled and randomized in a double blinded manner to receive either Artecom® or placebo (1:1 ratio) orally once a day for 3 consecutive days. All subjects will be evaluated for efficacy and safety for 28 days.

A second DSMB meeting and review of all available blinded safety data will occur after 191 participants have completed Day 28. A final DSMB meeting will be held after the completion of a study assessment by the last participant.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults age (≥19 years at the time of informed consent)
2. Body weight (≥ 45 kg at Screening)
3. Participants must be confirmed as having COVID-19 using real-time reverse transcription polymerase chain reaction (RT-PCR) test and specimens collected from upper airway (nasopharyngeal specimen) within 96 hours prior to randomization.
4. Females must be non-pregnant and non-lactating, and must use an acceptable, highly effective double contraception from Screening until study completion, including the follow-up period. Males must be surgically sterile (>30 days since vasectomy with no viable sperm), abstinent, or if engaged in sexual relations with a woman of childbearing potential (WOCBP), the participant and his partner must be surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or using an acceptable, highly effective contraceptive method from Screening until study completion, including the follow-up period.

   * Hormonal contraception (with approved oral contraceptives, long-acting implantable hormones, injectable hormones), intra uterine device, condoms , sterilization (vasectomy, tubal occlusion, etc.)

Exclusion Criteria:

1. Participants with clinically significant cardiovascular disease (including arrhythmia, corrected QT interval prolongation [QTcF> 470 msec for females, or >450 msec for males, at Screening])
2. Participants with clinically significant anemia (Hemoglobin <8.0 g/dL)
3. Participants who have hypersensitivity to main ingredients (pyronaridine tetraphosphate, artesunate) and any excipient in the IP
4. Participants who have gastrointestinal disease or surgical participant that may affect absorption, distribution, metabolism and excretion of drugs, current active gastritis, gastrointestinal /rectal bleeding, gastric ulcers, pancreatic abnormalities such as pancreatitis, etc. (simple appendectomy or hernia surgery not excluded)
5. Participants who have received antiviral drugs for the treatment of COVID-19 infection or other indications within 28 days prior to participation in the study or who have not had sufficient wash-out period of the antiviral drugs
6. Participants with severe renal impairment (estimated glomerular filtration rate ≤30 mL/min/1.73 m2)
7. Participants with severe hepatic impairment (Alanine aminotransferase or Aspartate aminotransferase ≥5x upper limit of normal) or have symptoms of abdominal pain or vomiting associated with Jaundice or Child-Pugh Stage B or C
8. Viral infections other than COVID-19 that requires administration of other antiviral agents (for example but not limited to human immunodeficiency virus, hepatitis B virus, hepatitis C virus)
9. Participants requiring mechanical ventilation (e.g. non-invasive ventilation, invasive mechanical ventilation, extracorporeal membrane oxygenation etc.). However, those who can be given oral administration are not exdluded.
10. Participants with chronic underlying diseases (such as uncontrolled diabetes, chronic kidney disease, chronic liver disease, chronic lung disease [including asthma, chronic obstructive pulmonary disease and tuberculosis], chronic cardiovascular disease, blood cancer, cancer participants with anti-cancer treatment, participants taking immunosuppressants, etc.), participants with high obesity (BMI > 40), dialysis participants, transplant participants whom are inadequate to participate in clinical trials based on the Investigator's discretion.
11. Pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study, including the follow-up period.
12. Participants who participated in another clinical trial / medical device clinical trial within 28 days from the date of signing the consent and received drug / operated medical device for clinical trial.
13. Participants who the Investigator has deemed inappropriate for inclusion in this study for any other reason.
14. Prior or ongoing medical conditions, medical history, physical findings, or laboratory abnormality that, in the Investigator's (or delegate's) opinion, could adversely affect the safety of the participant.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-04-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with clinical improvement as defined by an improvement of categories on the WHO Ordinal Scale of clinical status until Days 28. | follows up to 28 days
  * WHO Ordinal scale: 0. No clinical or virological evidence of infection
  1. No limitation of activities
  2. Limitation of activities
  3. Hospitalized, no oxygen therapy
  4. Oxygen by mask or nasal prongs
  5. Non-invasive ventilation or high-flow oxygen
  6. Intubation and mechanical ventilation
  7. Ventilation + additional organ support - Pressers, Renal replacement therapy (RRT), extracorporeal membrane oxygenation (ECMO)
  8. Death

SECONDARY OUTCOMES:
Time to clinical improvement was defined as time from randomization to an improvement of categories on the WHO Ordinal Scale of clinical status. | follows up to 28 days
  Clinical improvement within 28 days since start of treatment, defined as a decrease of at least 2 point from baseline of a nine-point WHO ordinal scale.
Changes in the WHO Ordinal Scale for Clinical Improvement until Days 28 compared to Baseline. | follows up to 28 days
  Compare statistical results of an increase or decrease in a nine-point WHO ordinal scale between two groups.
Changes in National Early Warning Score (NEWS) until Days 28 compared to Baseline. | follows up to 28 days
  NEWS determines the degree of illness of a patient and promotes critical care intervention. The score range from 0-20, with a higher score representing a higher risk of morbidity. Compare statistical results of an increase or decrease in NEWS between two groups.
Proportion of participants with negative for COVID-19 as determined by real-time RT-PCR test until Days 14. | follows up to 14 days
  Proportion of subjects who are RT-PCR negative for COVID-19
Changes in viral load until Days 14 compared to Baseline. | follows up to 14 days
  Viral load reduction of COVID-19 until Days 14 compared to the baseline.
The time to body temperature normalization after the administration of investigational Product (IP). | follows up to 28 days
  Maintaining underarm ≤36.7 °C, or oral ≤36.9°C, or rectal ≤37.3°C, or eardrum ≤37.2°C, for at least 24 hours without administering fever reducing medication after the administration of IP.
The time to respiratory rate normalization after the administration of IP. | follows up to 28 days
  Maintain 12/min ≤ respiratory rate ≤ 20/min for at least 24 hours.
The time to oxygen saturation (SpO2) normalization after the administration of IP. | follows up to 28 days
  SpO2 ≥95% for at least 24 hours.
Mortality rate at Day 28. | Day 28
  Compare the mortality rate between two groups.
Duration of hospitalization (Day 1 to Day 28). | follows up to 28 days
  Number of days the subject from the start of treatment to hospital discharge.
The incidence of adverse events (AEs). | follows up to 28 days
  The incidence rate of adverse events
The incidence of serious adverse events (SAEs). | follows up to 28 days
  The incidence rate of serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Belen L Dofitas, MD, PhD, Principal Investigator — Philippine General Hospital, University of the Philippines
Locations (4):
- Philippines (4):
  - De La Salle University Medical Center, Dasmariñas, Gov, D. Mangubat St, 4114 Cavite
  - The Medical City, Pasig, Ortigas Avenue, Barangay Ugong, Metro Manila
  - Lung Center of the Philippines, Quezon City, Quezon Avenue, Quezon City, 1100 Philippines
  - Philippine General Hospital, Manila, Taft Ave, Ermita, Manila, 1000 Metro

IPD SHARING:
Plan to Share IPD: No